CLINICAL TRIAL: NCT04034420
Title: SMART Family-Link Project: Capacity Building Online Platform for Training, Learning and Sharing (i-TLS) for Social and Service-related Workers
Brief Title: Capacity Building Online Platform for Social and Service-related Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UW 19-449
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-12

CONDITIONS: ICT
Keywords: Online platform; ICT; Family services

STUDY DESIGN:
Intervention Model Description: An online platform to provide training learning and sharing to social and service-related professionals for enhancing the quality of family services
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online training (Experimental): To receive self-paced online training and learning materials
  Interventions: Other: Online training platform

INTERVENTIONS:
Other: Online training platform — Self-paced training and learning materials in relation to family services

SUMMARY:
In the past few decades, Information and Communications Technology (ICT) have rapidly developed as effective, and probably the most cost-effective tools to connect most aspects of family lives. Alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also an increasing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes.

To gain more understanding of the potential new avenues of using ICT in programme implementation, The Hong Kong Jockey Club Charities Trust has initiated the Jockey Club SMART Family-Link Project in collaboration with The University of Hong Kong (HKU) and NGOs. This project aimed at helping 26 NGO-operated Integrated Family Service Centres and Integrated Service Centres (Centres), making effective use of information and communications technology (ICT) and data analytics, to enhance the quality and efficiency of their family service. Besides, it aims at building the capabilities of front-line workers so as to achieve the goal of enhancing family well-being by building an online training platform. We anticipated that the platform will benefit social workers or service-related workers in terms of knowledge transfer, experience sharing, and wisdom practice.

DETAILED DESCRIPTION:
In the past few decades, Information and Communications Technology (ICT) have rapidly developed as effective, and probably the most cost-effective tools to connect most, if not all, aspects of family lives. In Hong Kong, as of March 2016, the number of mobile service subscribers was 16.72 million, representing one of the highest penetration rates in the world at about 228.3 per cent; amongst these subscribers, 14.69 million were 3G/ 4G service customers and there is a surge to 20,557 Terabytes (or an average of 1,358 Megabytes per 2.5G/3G/4G mobile user) recorded for local mobile data usage, representing a growth of 1.18 times and 1.58 times over the same period in 2015 and 2014 respectively.

While alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also an increasing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes. It is believed that ICT helps facilitate access to interventions from a large variety of settings at all times, bringing the intervention to participants at times convenient to them and diminishing the influence of the situational constraints on intervention participation rates. The rise of ICT has created promising and potential new avenues and demand for implementing interventions related to mental health and parenting.

The Hong Kong Jockey Club Charities Trust has initiated the Jockey Club SMART Family-Link Project in collaboration with The University of Hong Kong (HKU) and NGOs, making effective use of information and communications technology (ICT) and data analytics, aimed at helping 26 NGO-operated Integrated Family Service Centres and Integrated Service Centres (Centres), to enhance the quality and efficiency of their family service. The project also aims at building the capabilities of front-line workers so as to achieve the goal of enhancing family well-being by building an online training platform.

The i-Training, Learning, and Sharing (i-TLS) platform will provide staff training and skills enhancing through carefully selected materials in one convenient location, forums for wisdom, experience, and information sharing between staff.

1. i-Training: Using a variety of computerized formats, the i-Training platform may bring professional training content to social workers at their convenience.
2. i-Learning: It provides a co-learning area for social and related service workers from different service centers to learn from and support each other, such as the NGO-shared best practice and the updated ICT information in relation to family services and activities. This may enhance service effectiveness.
3. i-Sharing: It provides social and service-related workers with an instant online means to share experiences and have discussions

The Platform will benefit social workers or service-related workers in terms of knowledge transfer, experience sharing, and wisdom practice.

The goal of the study is to assess the feasibility and effectiveness of using online i-TLS platform to provide training and encourage a co-learning and sharing culture amongst social work professionals.

A process evaluation will be performed to evaluate the process of each component of the program. Qualitative and quantitative assessments will be used to evaluate the effectiveness of the activities

ELIGIBILITY:
Inclusion Criteria:

* Social service stakeholders (including social workers, service-related workers)
* Chinese speaking
* Able to complete the questionnaire

Exclusion Criteria:

* Subjects who fail to meet the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction on the online i-TLS platform and its content | immediately after using the platform
  Outcome based questions will be used to assess participants' satisfaction level on using the i-TLS platform and its content. The higher score indicates the better outcome.

SECONDARY OUTCOMES:
The perceived usefulness of training platform and its materials | 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Outcome based questions will be used to assess the perceived usefulness of training platform and its information.
The perceived usefulness of learning platform and its materials | 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Outcome based questions will be used to assess the perceived usefulness of learning platform and its information
The perceived usefulness of sharing forum | 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  Outcome based questions will be used to assess the perceived usefulness of sharing forum

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: i-Training, Learning, Sharing (i-TLS) platform — https://i-tls.jcsfl.hk/